CLINICAL TRIAL: NCT00729495
Title: Phase I, Randomized, Open-Label, 2-Way Crossover Study to Evaluate Relative Bioavailability of Single Oral Dose of Celecoxib Administered as Marketed Product, or Overencapsulated Capsule in Healthy Volunteers
Brief Title: Phase I Study to Evaluate Bioavailability of Overencapsulated Celecoxib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POZEN (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Mark Sostek, MD, Medical Science Director, Development Project, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: D1120C00007
Record Dates: First submitted 2008-08-05; First posted 2008-08-07 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Healthy Volunteer
Keywords: Phase I,; Healthy; Volunteer; Study
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): marketed celecoxib
  Interventions: Drug: celecoxib
- 2 (Experimental): overencapsulated celecoxib
  Interventions: Drug: celecoxib

INTERVENTIONS:
Drug: celecoxib — dose form
  Other Names: Celebrex

SUMMARY:
Phase I study designed to test the hypothesis that overencapsulated celecoxib 200 mg qd is bioequivalent to commercial celecoxib 200 mg qd. Approximately 90 healthy volunteers will be randomized to yield approximately 80 completers. The study is an open label, randomized, 2-way crossover with single dosing followed by a 7-day washout period between treatment arms

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects 18-55 yrs. of age (inclusive) at Screening Visit
* Body Mass Index (BMI) of greater than or equal to 19 to less than or equal to 30 kg/m2 and weight of greater than or equal to 50 to less than or equal to 100 kg
* Clinically normal physical exams and laboratory measurements

Exclusion Criteria:

* Subject has received another investigational drug within 4 weeks preceeding this study or planning to participate in another study at any time during the period of this study
* Any significant medical or psychiatric condition that could affect the interpretation of the PK data, or which otherwise would contraindicate participation in a clinical trial
* Any GI disease, abnormality or gastric surgery that may interfere with gastric emptying, motility and drug absorption
* Subject who has donated a unit of blood or plasma within 3 months prior to the Screening Visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | pre-dose, baseline and multiple times post-dose

SECONDARY OUTCOMES:
Safety | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, MD, Study Director — AstraZeneca; Christopher Billings, DO, Principal Investigator — Bio-Kinetic Clinical Applications, LLC
Locations (1):
- Research, Springfield, Missouri, United States